CLINICAL TRIAL: NCT03345914
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Dupilumab Administered Concomitantly With Topical Corticosteroids in Patients, ≥6 Years to <12 Years of Age, With Severe Atopic Dermatitis
Brief Title: Study to Investigate the Efficacy and Safety of Dupilumab Administered With Topical Corticosteroids (TCS) in Participants ≥6 to <12 Years With Severe Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-AD-1652; 2016-004997-16 (EudraCT Number)
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Dermatitis, Atopic
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive dupilumab, dosing regimen 1
  Interventions: Drug: Dupilumab; Other: Background Treatment: Topical Corticosteroids; Other: Background Treatment: Moisturizers
- Group 2 (Experimental): Participants will receive dupilumab, dosing regimen 2
  Interventions: Drug: Dupilumab; Other: Background Treatment: Topical Corticosteroids; Other: Background Treatment: Moisturizers
- Group 3 (Experimental): Participants will receive matching placebo
  Interventions: Drug: Matching Placebo; Other: Background Treatment: Topical Corticosteroids; Other: Background Treatment: Moisturizers

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form: Solution for injection in pre-filled syringe;
  Route of administration: Subcutaneous (SC)
  Other Names: DUPIXENT®; REGN668; SAR231893
  Arms: Group 1; Group 2
Drug: Matching Placebo — Pharmaceutical form: Solution for injection;
  Route of administration: Subcutaneous (SC)
  Arms: Group 3
Other: Background Treatment: Topical Corticosteroids — All participants are required to initiate treatment with a medium potency TCS using a standardized regimen. It is recommended that participants use triamcinolone acetonide 0.1% cream, fluocinolone acetonide 0.025% cream, or clobetasone butyrate 0.05%.
Other: Background Treatment: Moisturizers — All participants should apply moisturizers throughout the study. All types of moisturizers are permitted, but participants may not initiate treatment with prescription moisturizers. Participants may continue using stable doses of such moisturizers if initiated before the screening visit.

SUMMARY:
The main objective of the trial is to demonstrate the efficacy of dupilumab administered concomitantly with topical corticosteroids (TCS) in participants ≥6 years to <12 years of age with severe atopic dermatitis (AD).

The secondary objective is to assess the safety of dupilumab administered concomitantly with TCS in patients ≥6 years to <12 years of age with severe AD.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of AD according to the American Academy of Dermatology consensus criteria (Eichenfield 2003) at screening visit
2. Chronic AD diagnosed at least 1 year prior to the screening visit
3. IGA = 4 at screening and baseline visits
4. EASI ≥21 at the screening and baseline visits
5. BSA ≥15% at screening and baseline visits
6. Documented recent history (within 6 months before the baseline visit) of inadequate response to topical AD medication(s)
7. At least 11 (of a total of 14) applications of a stable dose of topical emollient (moisturizer) twice daily during the 7 consecutive days immediately before the baseline visit

Key Exclusion Criteria:

1. Participation in a prior dupilumab clinical study
2. Treatment with a systemic investigational drug before the baseline visit
3. Treatment with a topical investigational drug within 2 weeks prior to the baseline visit
4. Treatment with crisabarole within 2 weeks prior to the baseline visit
5. History of important side effects of medium potency topical corticosteroids (e.g, intolerance to treatment, hypersensitivity reactions, significant skin atrophy, systemic effects), as assessed by the investigator or patient's treating physician
6. Treatment with a topical calcineurin inhibitor (TCI) within 2 weeks prior to the baseline visit
7. Having used any of the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during the first 4 weeks of study treatment:

   1. Immunosuppressive/immunomodulating drugs (e.g, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon gamma, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
   2. Phototherapy for AD
8. Treatment with biologics, as follows:

   1. Any cell-depleting agents including but not limited to rituximab:

      within 6 months before the baseline visit, or until lymphocyte and CD 19+ lymphocyte count returns to normal, whichever is longer
   2. Other biologics: within 5 half-lives (if known) or 16 weeks before the baseline visit, whichever is longer
9. Treatment with a live (attenuated) vaccine within 4 weeks before the baseline visit
10. Body weight <15 kg at baseline

Note: Other Inclusion/ Exclusion criteria apply

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 367 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (56):
- United States (30):
  - Regeneron Research Site, Birmingham, Alabama
  - Regeneron Research Site, Gilbert, Arizona
  - Regeneron Research Site, Bakersfield, California
  - Regeneron Research Site, Long Beach, California
  - Regeneron Research Site, Mission Viejo, California
  - Regeneron Research Site, Rolling Hills Estates, California
  - Regeneron Research Site, San Diego, California
  - Regeneron Research Site, Denver, Colorado
  - Regeneron Research Site, Coral Gables, Florida
  - Regeneron Research Site, Tampa, Florida
  - Regeneron Research Site, Macon, Georgia
  - Regeneron Research Site, Sandy Springs, Georgia
  - Regeneron Research Site, Chicago, Illinois
  - Regeneron Research Site, Normal, Illinois
  - Regeneron Research Site, Rockville, Maryland
  - Regeneron Research Site, Ypsilanti, Michigan
  - Regeneron Research Site, Minneapolis, Minnesota
  - Regeneron Research Site, St Louis, Missouri
  - Regeneron Research Site, Forest Hills, New York
  - Regeneron Research Site, New York, New York
  - Regeneron Research Site, Rochester, New York
  - Regeneron Research Site, Gahanna, Ohio
  - Regeneron Research Site, Portland, Oregon
  - Regeneron Research Site, Philadelphia, Pennsylvania
  - Regeneron Research Site, Charleston, South Carolina
  - Regeneron Research Site, North Charleston, South Carolina
  - Regeneron Research Site, Bellaire, Texas
  - Regeneron Research Site, San Antonio, Texas
  - Regeneron Research Site, Norfolk, Virginia
  - Regeneron Research Site, Seattle, Washington
- Canada (4):
  - Regeneron Research Site, Calgary, Alberta
  - Regeneron Research Site, Markham, Ontario
  - Regeneron Research Site, Peterborough, Ontario
  - Regeneron Research Site, Montreal, Quebec
- Czechia (2):
  - Regeneron Research Site, Kutná Hora
  - Regeneron Research Site, Ústí nad Labem
- Germany (7):
  - Regeneron Research Site, Munich, Bavaria
  - Regeneron Research Site, Osnabrück, Lower Saxony
  - Regeneron Research Site, Münster, North Rhine-Westphalia
  - Regeneron Research Site, Dresden, Saxony
  - Regeneron Research Site, Gera, Thuringia
  - Regeneron Research Site, Bad Bentheim
  - Regeneron Research Site, Hamburg
- Poland (9):
  - Regeneron Research Site, Wroclaw, Lower Silesian Voivodeship
  - Regeneron Research Site, Krakow, Malopolska
  - Regeneron Research Site, Bialystok
  - Regeneron Research Site, Bydgoszcz
  - Regeneron Research Site, Gdansk
  - Regeneron Research Site, Katowice
  - Regeneron Research Site, Lodz
  - Regeneron Research Site, Świętokrzyskie
  - Regeneron Research Site, Warsaw
- United Kingdom (4):
  - Regeneron Research Site, London
  - Regeneron Research Site, Manchester
  - Regeneron Research Site, Newcastle upon Tyne
  - Regeneron Research Site, Sheffield

REFERENCES:
- [Derived] Langley RG, Gherardi G, Coleman A, Ardeleanu M, Rodriguez-Marco A, Levy S, Bansal A, Chen Z, Rossi AB, Shumel B, Khokhar FA. The Safety Data of Dupilumab for the Treatment of Moderate-to-Severe Atopic Dermatitis in Infants, Children, Adolescents, and Adults. Am J Clin Dermatol. 2025 Nov;26(6):981-1002. doi: 10.1007/s40257-025-00952-w. Epub 2025 Sep 24. PMID 40993471
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Cork MJ, Thaci D, Eichenfield LF, Arkwright PD, Chen Z, Thomas RB, Kosloski MP, Dubost-Brama A, Prescilla R, Bansal A, Levit NA. Dupilumab Safety and Efficacy in a Phase III Open-Label Extension Trial in Children 6-11 Years of Age with Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2023 Nov;13(11):2697-2719. doi: 10.1007/s13555-023-01016-9. Epub 2023 Sep 26. PMID 37750994
- [Derived] Siegfried EC, Cork MJ, Katoh N, Zhang H, Chuang CC, Thomas RB, Rossi AB, Cyr SL, Zhang A. Dupilumab Provides Clinically Meaningful Responses in Children Aged 6-11 Years with Severe Atopic Dermatitis: Post Hoc Analysis Results from a Phase III Trial. Am J Clin Dermatol. 2023 Sep;24(5):787-798. doi: 10.1007/s40257-023-00791-7. Epub 2023 Jun 10. PMID 37300760
- [Derived] Paller AS, Yosipovitch G, Weidinger S, DiBenedetti D, Whalley D, Gadkari A, Guillemin I, Zhang H, Eckert L, Chao J, Bansal A, Chuang CC, Delevry D. Development, Psychometric Validation and Responder Definition of Worst Itch Scale in Children with Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2022 Dec;12(12):2839-2850. doi: 10.1007/s13555-022-00804-z. Epub 2022 Oct 21. PMID 36269504
- [Derived] Paller AS, Wollenberg A, Siegfried E, Thaci D, Cork MJ, Arkwright PD, Gooderham M, Sun X, O'Malley JT, Khokhar FA, Vakil J, Bansal A, Rosner K, Shumel B, Levit NA. Laboratory Safety of Dupilumab in Patients Aged 6-11 Years with Severe Atopic Dermatitis: Results from a Phase III Clinical Trial. Paediatr Drugs. 2021 Sep;23(5):515-527. doi: 10.1007/s40272-021-00459-x. Epub 2021 Aug 31. PMID 34462864
- [Derived] Simpson EL, Paller AS, Siegfried EC, Thaci D, Wollenberg A, Cork MJ, Marcoux D, Huang R, Chen Z, Rossi AB, Shumel B, Sierka D, Bansal A. Dupilumab Demonstrates Rapid and Consistent Improvement in Extent and Signs of Atopic Dermatitis Across All Anatomical Regions in Pediatric Patients 6 Years of Age and Older. Dermatol Ther (Heidelb). 2021 Oct;11(5):1643-1656. doi: 10.1007/s13555-021-00568-y. Epub 2021 Aug 24. PMID 34427891
- [Derived] Kamal MA, Kovalenko P, Kosloski MP, Srinivasan K, Zhang Y, Rajadhyaksha M, Lai CH, Kanamaluru V, Xu C, Sun X, Simpson EL, Paller AS, Siegfried EC, Shumel B, Bansal A, Al-Huniti N, Davis JD. The Posology of Dupilumab in Pediatric Patients With Atopic Dermatitis. Clin Pharmacol Ther. 2021 Nov;110(5):1318-1328. doi: 10.1002/cpt.2366. Epub 2021 Aug 24. PMID 34270797
- [Derived] Simpson EL, de Bruin-Weller M, Bansal A, Chen Z, Nelson L, Whalley D, Prescilla R, Guillemin I, Delevry D. Definition of Clinically Meaningful Within-Patient Changes in POEM and CDLQI in Children 6 to 11 Years of Age with Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2021 Aug;11(4):1415-1422. doi: 10.1007/s13555-021-00543-7. Epub 2021 May 27. PMID 34046851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 474 participants were screened for study eligibility at multiple sites in the United States and Europe. Screen failure was mostly due to inclusion/exclusion criteria not met and "other" reasons. The majority of participants (221/367) were enrolled at study sites in the United States.
Pre-assignment Details: A total of 474 participants were screened. 367 participants randomized in 1:1:1 ratio to 1 of 3 treatment groups. 5 randomized participants were not treated (2 in placebo + TCS group & 3 in combined dupilumab + TCS group). Participants randomized to receive Dupilumab 100 mg or 200 mg Q2W + TCS, Dupilumab 300 mg Q4W + TCS or matching placebo.
Groups:
- Placebo + TCS: Participants received matching placebo every 2 weeks (Q2W) or every 4 weeks (Q4W) during the 16-week double-blind treatment phase. Matching placebo was administered concomitantly with topical corticosteroids (TCS), including doubling the amount of placebo on Day 1 to match the loading dose.
- Dupilumab 300 mg Q4W + TCS: Participants received subcutaneous injections of 600 milligrams (mg) loading dose on Day 1, then 300 mg of Dupilumab every 4 weeks (Q4W) from Week 4 to Week 12. Topical corticosteroids (TCS) were administered concomitantly during the 16-week double-blind treatment phase.
- Dupilumab 100 mg or 200 mg Q2W + TCS: Participants received subcutaneous injections of 100 milligrams (mg) or 200 mg of Dupilumab every 2 weeks (Q2W). For 100 mg Q2W treatment group, participants received a 200 mg loading dose on Day 1, then 100 mg Q2W from Week 2 to Week 14. For 200 mg Q2W treatment group, participants received a 400 mg loading dose on Day 1, then 200 mg Q2W from Week 2 to Week 14. Topical corticosteroids (TCS) were administered concomitantly in all groups during the 16-week double-blind treatment phase.
Period: Overall Study
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Started | 123 | 122 | 122
Completed Week 16 Study Treatment | 114 | 118 | 119
Completed Week 28 End of Study | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 123 | 122 | 122
Not completed — Transition to another study at week 16 | 80 | 86 | 78
Not completed — Transition to OLE during follow-up | 37 | 33 | 39
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 2
Not completed — Other | 1 | 1 | 1
Not completed — Ongoing | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS | Total
Number analyzed (Participants) | 123 | 122 | 122 | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (1.76) | 8.5 (1.74) | 8.5 (1.68) | 8.5 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 65 | 57 | 184
  Male | 61 | 57 | 65 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 16 | 16 | 45
  Not Hispanic or Latino | 110 | 106 | 106 | 322
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 5 | 10 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 19 | 20 | 62
  White | 77 | 89 | 88 | 254
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 9 | 4 | 23
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: Score on a Scale] — The EASI assesses severity and extent of atopic dermatitis. Scores range from 0-72. Four AD disease characteristics (erythema, thickness, scratching, and lichenification) are assessed for severity on a scale of "0" (absent) through "3" (severe). Area of involvement assessed as a percentage by body area of head, trunk, upper limbs and lower limbs and converted to a score of 0 to 6. Higher score indicates increased extent and severity of atopic dermatitis.
  Score on a Scale | 39.0 (12.01) | 37.4 (12.45) | 37.3 (10.86) | 37.9 (11.79)
Investigator's Global Assessment (IGA) Score [Mean (Standard Deviation); unit: Score on a Scale] — IGA is an assessment instrument used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Score on a Scale | 4.0 (0.00) | 4.0 (0.09) | 4.0 (0.00) | 4.0 (0.05)
Weekly Average of Daily Worst Itch Score [Mean (Standard Deviation); unit: Score on a Scale] — The worst itch scale is a simple assessment tool that participants will use to report the intensity of their pruritus (itch). This is an 11-point scale (0 to 10) in which 0 indicates no itching while 10 indicates worst itching possible. Participants will be asked to answer 2 questions daily throughout the entire study (screening period, treatment period, and follow-up period). The daily worst itch score will be calculated as the worse of the scores for the 2 questions. Population: Here "number analyzed" represents the number of participants who were evaluable for this measure.
  Score on a Scale
    number analyzed (Participants) | 123 | 122 | 120 | 365
    (all) | 7.7 (1.54) | 7.8 (1.58) | 7.8 (1.52) | 7.8 (1.54)
Body Surface Area (BSA) of Atopic Dermatitis [Mean (Standard Deviation); unit: Percentage of BSA] — BSA affected by AD will be assessed for each section of the body using the rule of nines (the possible highest score for each region is: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and will be reported as a percentage of all major body sections combined. The proportion assigned to different body regions is different in younger children as compared to older children (head and neck area is assigned a higher proportion in younger children as compared to older children).
  Percentage of BSA | 60.2 (21.46) | 54.8 (21.58) | 57.8 (20.04) | 57.6 (21.10)
SCORing Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: Score on a Scale] — SCORAD is used to assess the extent and severity of AD. Extent and severity of eczema as well as subjective symptoms (insomnia, etc) were assessed and scored. SCORAD total score range is from 0 (absent disease) to 103 (severe disease).
  Score on a Scale | 72.9 (12.01) | 75.6 (11.71) | 72.3 (10.83) | 73.6 (11.59)
Patient Oriented Eczema Measure (POEM) [Mean (Standard Deviation); unit: Score on a Scale] — POEM is a 7-item, validated questionnaire used to assess disease symptoms in children and adults. The format is a response to 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on frequency of these disease symptoms during the past week (ie, 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days) with a scoring system of 0 to 28; the total score reflects disease-related morbidity. A high score is indicative of a poor quality of life.
  Score on a Scale | 20.7 (5.48) | 21.3 (5.51) | 20.5 (5.50) | 20.9 (5.49)
Children's Dermatology Life Quality Index (CDLQI) Total Score [Mean (Standard Deviation); unit: Score on a Scale] — CDLQI is a validated 10 question tool to measure the impact of skin disease on quality of life (QOL) in children by assessing how much the skin problem has affected the participant over the past week. Nine questions are scored as follows: Very much = 3, Quite a lot = 2, Only a little = 1, Not at all or unanswered = 0. Question 7 has added possible response, which is scored as 3. CDLQI equals the sum of the score of each question (maximum = 30, minimum = 0). Higher the score, the greater the impact on QOL. Data presented reflects the mean & standard deviation of the CDLQI total scores.
  Score on a Scale | 14.6 (7.41) | 16.2 (7.85) | 14.5 (6.78) | 15.1 (7.38)
Dermatitis Family Index (DFI) [Mean (Standard Deviation); unit: Score on a Scale] — DFI is a 10-item questionnaire with items inquiring about housework, food preparation, sleep, family leisure activity, shopping, expenditure, tiredness, emotional distress, relationships and the impact of helping with treatment on the primary caregiver's life. The DFI questions are scored on a four-point Likert scale ranging from 0 to 3, so that the total DFI score ranges from 0 to 30. Timeframe of reference is the past week. A higher DFI score indicates greater impairment in family QOL as affected by atopic dermatitis.
  Score on a Scale | 15.0 (7.54) | 16.9 (8.65) | 14.9 (7.05) | 15.6 (7.81)
Patient Reported Outcomes Measurements Information Systems (PROMIS) Anxiety Scale [Mean (Standard Deviation); unit: Score on a Scale] — PROMIS Anxiety instrument measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), & somatic symptoms related to arousal (racing heart, dizziness). Each question has 5 response options ranging in value from 1-5 (1=Never, 2=Almost never, 3=Sometimes, 4=Often, 5=Almost Always). For an 8-item form, lowest possible total raw score is 8; highest possible total raw score is 40. For a 6-item form, lowest possible total raw score is 6; highest possible total raw score is 30. Higher score indicates greater severity of symptoms. Population: Here number analyzed represents the number of participants who were evaluable for this measure.
  Score on a Scale
    number analyzed (Participants) | 121 | 121 | 121 | 363
    (all) | 57.3 (11.62) | 59.8 (13.66) | 58.6 (11.32) | 58.6 (12.25)
Patient Reported Outcomes Measurements Information Systems (PROMIS) Depression Scale [Mean (Standard Deviation); unit: Score on a Scale] — PROMIS Depression instrument assesses self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness) & social cognition (loneliness, interpersonal alienation), & decreased positive affect & engagement (loss of interest, meaning & purpose). Each question has 5 response options ranging in value from 1-5 (1=Never, 2=Almost never, 3=Sometimes, 4=Often, 5= Almost Always). For 8-item form, lowest possible total raw score is 8 and highest is 40. For 6-item form, lowest possible total raw score is 6 and highest is 30. Higher score indicates greater severity of symptoms. Population: Here number analyzed represents the number of participants who were evaluable for this measure.
  Score on a Scale
    number analyzed (Participants) | 121 | 121 | 121 | 363
    (all) | 55.0 (12.05) | 58.1 (12.77) | 56.3 (11.22) | 56.4 (12.06)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) 0 or 1 at Week 16
Description: The IGA was an assessment instrument used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe). The full analysis set (FAS) included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Values after first rescue treatment used were set to missing. Participants with missing score at Week 16 were considered as a non-responder.
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percentage of Participants | 11.4 | 32.8 | 29.5
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; A 2-sided hierarchical testing procedure was used for the primary and secondary endpoints in a pre-specified order. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — The Cochran-Mantel-Haenszel (CMH) test adjusted by randomization strata (baseline weight group (< 30 kilograms (kg) or ≥ 30 kg) and region (North America or Europe) was used for the analysis of percentage of participants with IGA 0 or 1 at Week 16; Percentage difference = 18.1, 95% CI 2-sided [8.28 to 27.97]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — The Cochran-Mantel-Haenszel (CMH) test adjusted by randomization strata (baseline weight group (< 30 kg or ≥ 30 kg) and region (North America or Europe) was used for the analysis of percentage of participants with IGA 0 or 1 at Week 16; Percentage difference = 21.4, 95% CI 2-sided [11.36 to 31.45]

2. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index -75 (EASI-75) (≥ 75 Percent (%) Improvement From Baseline) at Week 16
Description: The EASI assesses severity and extent of atopic dermatitis (AD). Scores range from 0-72. Four AD disease characteristics (erythema, thickness, scratching, and lichenification) were assessed for severity on a scale of "0" (absent) through "3" (severe). Area of involvement assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Values after first rescue treatment used were set to missing. Participants with missing score at week 16 were considered as a non-responder.
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percentage of Participants | 26.8 | 69.7 | 67.2
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — The Cochran-Mantel-Haenszel (CMH) test adjusted by randomization strata (baseline weight group (< 30 kg or ≥ 30 kg) and region (North America or Europe) was used for the analysis of percentage of participants with EASI-75 at Week 16; Percentage difference = 40.4, 95% CI 2-sided [28.95 to 51.82]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Percentage difference = 42.8, 95% CI 2-sided [31.54 to 54.15]

3. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 16
Description: The EASI assesses severity and extent of AD. Scores range from 0-72. Four AD disease characteristics (erythema, thickness, scratching, and lichenification) were assessed for severity on a scale of "0" (absent) through "3" (severe). Area of involvement assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Time Frame: Baseline (Day 1), Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percent change | -48.6 (2.46) [lower limit 2.46] | -82.1 (2.37) [lower limit 2.37] | -78.4 (2.35) [lower limit 2.35]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — The confidence interval (CI) with p-value was based on treatment difference (Dupilumab group vs placebo) of the LS mean percent change using ANCOVA model with baseline measurement as covariate and the treatment, randomization strata as fixed factors; Least Square Mean Difference = -29.8, 95% CI 2-sided [-36.33 to -23.24]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -33.4, 95% CI 2-sided [-40.06 to -26.82]

4. Secondary Outcome: Percent Change From Baseline in Weekly Average of Daily Worst Itch Score at Week 16
Description: The worst itch scale was a simple assessment tool that participants used to report the intensity of their pruritus (itch). This was an 11-point scale (0 to 10) in which 0 indicated no itching while 10 indicated worst itching possible. Participants were asked to answer 2 questions daily throughout the entire study (screening period, treatment period, and follow-up period). The daily worst itch score was calculated as the worse of the scores for the 2 questions. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Time Frame: Baseline (Day 1), Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percent change | -25.9 (2.90) [lower limit 2.90] | -54.6 (2.89) [lower limit 2.89] | -57.0 (2.77) [lower limit 2.77]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -31, 95% CI 2-sided [-38.76 to -23.26]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -28.6, 95% CI 2-sided [-36.47 to -20.82]

5. Secondary Outcome: Percentage of Participants With Improvement (Reduction From Baseline) of Weekly Average of Daily Worst Itch Score ≥3 Points at Week 16
Description: The worst itch scale was a simple assessment tool that participants used to report the intensity of their pruritus (itch). This was an 11-point scale (0 to 10) in which 0 indicated no itching while 10 indicated worst itching possible. Participants were asked to answer 2 questions daily throughout the entire study (screening period, treatment period, and follow-up period). The daily worst itch score was calculated as the worse of the scores for the 2 questions. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Values after first rescue treatment used were set to missing. Participants with missing score at week 16 were considered as a non-responder. Here "Number of participants analyzed" = number of participants who were evaluated for this specific endpoint.
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 121 | 120
Percentage of Participants | 21.1 | 60.3 | 67.5
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-values were derived by Cochran-Mantel-Haenszel (CMH) test stratified by region [North America vs Europe] and baseline weight group [< 30 kg vs ≥ 30 kg]; Percentage difference = 46.4, 95% CI 2-sided [35.3 to 57.42]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage difference = 39.2, 95% CI 2-sided [27.88 to 50.51]

6. Secondary Outcome: Percentage of Participants With Improvement (Reduction From Baseline) of Weekly Average of Daily Worst Itch Score ≥4 Points at Week 16
Description: as for outcome 5
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 122 | 120 | 120
Percentage of Participants | 12.3 | 50.8 | 58.3
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage difference = 46, 95% CI 2-sided [35.47 to 56.61]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage difference = 38.5, 95% CI 2-sided [27.86 to 49.21]

7. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index - 50 (EASI-50) (≥ 50% Improvement From Baseline) at Week 16
Description: The EASI assessed severity and extent of AD. Scores range from 0-72. Four AD disease characteristics (erythema, thickness, scratching, and lichenification) were assessed for severity on a scale of "0" (absent) through "3" (severe). Area of involvement assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Values after first rescue treatment used were set to missing. Participants with missing score at week 16 were considered as a non-responder.
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percentage of Participants | 43.1 | 91.0 | 82.8
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage difference = 39.7, 95% CI 2-sided [28.68 to 50.72]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage difference = 47.9, 95% CI 2-sided [37.77 to 58.01]

8. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index - 90 (EASI - 90) (≥ 90% Improvement From Baseline) at Week 16
Description: The EASI assessed the severity and extent of atopic dermatitis (AD). Scores range from 0-72. Four AD disease characteristics (erythema, thickness, scratching, and lichenification) were assessed for severity on a scale of "0" (absent) through "3" (severe). Area of involvement assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Values after first rescue treatment used were set to missing. Participants with missing score at week 16 were considered as a non-responder.
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percentage of Participants | 7.3 | 41.8 | 30.3
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage difference = 23, 95% CI 2-sided [13.65 to 32.38]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage difference = 34.5, 95% CI 2-sided [24.6 to 44.37]

9. Secondary Outcome: Time to Achieve ≥ 4 Point Reduction of Weekly Average of Daily Worst Itch Score From Baseline During the 16-week Treatment Period
Description: The worst itch scale: simple assessment tool that participants used to report intensity of their pruritus (itch). This was an 11-point scale (0 to 10) where 0 (no itching) and 10 (worst itching) possible. Participants were asked to answer 2 questions daily throughout the entire study (screening period, treatment period, & follow-up period). The daily worst itch score was calculated as worse of scores for 2 questions. FAS was used. Time to event is calculated in weeks as (date of first event - date of first dose)/7. The event of NRS reduction ≥ 4 was based on observed data without setting data to be non-responder after rescue treatment use. Here "Number of participants analyzed" = number of participants who were evaluated for this specific endpoint & "NA" represents "Not computable" as only 12.3% of participants achieved NRS reduction during 16-week treatment period & hence median time to achieve ≥ 4-point reduction of NRS for placebo +TCS treated participants could not be reported.
Time Frame: Baseline (Day 1) up to Week 16
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 122 | 120 | 120
Weeks | NA [NA to NA] — NA represents "Not computable" as only 12.3% of participants achieved NRS reduction during 16-week treatment period & hence median time to achieve ≥ 4-point reduction of NRS for placebo +TCS treated participants could not be reported. | 10.0 [7 to 13] | 10.0 [8 to 12]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cox model — [p-value comment as in outcome 5, analysis 1]; Hazard ratios = 3.114, 95% CI 2-sided [2.097 to 4.624]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cox model — [p-value comment as in outcome 5, analysis 1]; Hazard ratios = 2.921, 95% CI 2-sided [1.957 to 4.36]

10. Secondary Outcome: Time to Achieve ≥ 3 Point Reduction of Weekly Average of Daily Worst Itch Score From Baseline During the 16-week Treatment Period
Description: The worst itch scale: a simple assessment tool that participants used to report intensity of their pruritus (itch). This was an 11-point scale (0 to 10) where 0 (no itching) & 10 (worst itching) possible. Participants were asked to answer 2 questions daily throughout the entire study (screening period, treatment period, & follow-up period). Daily worst itch score was calculated as worse of scores for 2 questions. FAS was used. Time to event is calculated in weeks as (date of first event - date of first dose)/7. The event of NRS reduction ≥ 3 was based on observed data without setting data to be non-responder after rescue treatment use. Here "Number of participants analyzed" = number of participants who were evaluated for this specific endpoint & "NA" represents "Not computable" as only 21.1% of participants achieved NRS reduction during 16-week treatment period & hence median time to achieve ≥ 3-point reduction of NRS for placebo +TCS treated participants could not be reported.
Time Frame: Baseline (Day 1) up to Week 16
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 121 | 120
Weeks | NA [11 to NA] — NA represents "Not computable" as only 21.1% of participants achieved NRS reduction during 16-week treatment period & hence median time to achieve ≥ 3-point reduction of NRS for placebo +TCS treated participants could not be reported. | 6.0 [5 to 9] | 5.0 [5 to 7]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cox model — [p-value comment as in outcome 5, analysis 1]; Hazard ratios = 2.278, 95% CI 2-sided [1.631 to 3.182]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cox model — [p-value comment as in outcome 5, analysis 1]; Hazard ratios = 2.075, 95% CI 2-sided [1.481 to 2.908]

11. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Affected by Atopic Dermatitis (AD) at Week 16
Description: BSA affected by AD was assessed for each section of the body using the rule of nines (the possible highest score for each region is: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and were reported as a percentage of all major body sections combined. The proportion assigned to different body regions were different in younger children as compared to older children (head and neck area is assigned a higher proportion in younger children as compared to older children). The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Time Frame: Baseline (Day 1), Week 16
Measure: Least Squares Mean (Standard Error); unit: Percentage of BSA
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percentage of BSA | -21.65 (1.721) [lower limit 1.721] | -40.53 (1.648) [lower limit 1.648] | -39.37 (1.629) [lower limit 1.629]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -17.72, 95% CI 2-sided [-22.272 to -13.161]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -18.88, 95% CI 2-sided [-23.479 to -14.289]

12. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) at Week 16
Description: SCORAD was used to assess the extent and severity of AD. Extent and severity of eczema as well as subjective symptoms (insomnia, etc) were assessed and scored. SCORAD total score ranges from 0 (absent disease) to 103 (severe disease). The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Time Frame: Baseline (Day 1), Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percent change | -29.8 (2.26) [lower limit 2.26] | -62.4 (2.13) [lower limit 2.13] | -60.2 (2.11) [lower limit 2.11]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -30.4, 95% CI 2-sided [-36.3 to -24.48]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -32.6, 95% CI 2-sided [-38.57 to -26.59]

13. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) at Week 16
Description: CDLQI was a validated 10 question tool to measure the impact of skin disease on the quality of life (QOL) in children by assessing how much the skin problem has affected the participant over the past week. Nine questions were scored as follows: Very much = 3, Quite a lot = 2, Only a little = 1, Not at all or unanswered = 0. Question 7 has an added possible response, which was scored as 3. CDLQI equals the sum of the score of each question (maximum = 30, minimum = 0). Higher the score, the greater the impact on QOL. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Data presented reflects the mean & standard deviation of the CDLQI total scores.
Time Frame: Baseline (Day 1), Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Score on a Scale | -6.4 (0.51) [lower limit 0.51] | -10.6 (0.47) [lower limit 0.47] | -10.7 (0.46) [lower limit 0.46]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -4.3, 95% CI 2-sided [-5.62 to -2.99]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -4.2, 95% CI 2-sided [-5.57 to -2.89]

14. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) at Week 16
Description: POEM was a 7-item, validated questionnaire used to assess disease symptoms in children and adults. The format was a response to 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on frequency of these disease symptoms during the past week (ie, 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days) with a scoring system of 0 to 28; the total score reflected the disease-related morbidity. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). A high score is indicative of a poor quality of life.
Time Frame: Baseline (Day 1), Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Score on a Scale | -5.3 (0.69) [lower limit 0.69] | -13.6 (0.65) [lower limit 0.65] | -13.4 (0.65) [lower limit 0.65]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -8.1, 95% CI 2-sided [-9.96 to -6.31]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -8.3, 95% CI 2-sided [-10.13 to -6.43]

15. Secondary Outcome: Change From Baseline in Weekly Average of Daily Worst Itch Score at Week 16
Description: as for outcome 4
Time Frame: Baseline (Day 1), Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Score on a Scale | -2.05 (0.215) [lower limit 0.215] | -4.22 (0.207) [lower limit 0.207] | -4.45 (0.206) [lower limit 0.206]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -2.41, 95% CI 2-sided [-2.984 to -1.831]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -2.18, 95% CI 2-sided [-2.754 to -1.599]

16. Secondary Outcome: Change From Baseline in Dermatitis Family Index (DFI) at Week 16
Description: DFI was a 10-item questionnaire with items inquiring about housework, food preparation, sleep, family leisure activity, shopping, expenditure, tiredness, emotional distress, relationships and the impact of helping with treatment on the primary caregiver's life. The DFI questions were scored on a four-point Likert scale ranging from 0 to 3, so that the total DFI score ranges from 0 to 30. Timeframe of reference was the past week. A higher DFI score indicated greater impairment in family Quality of life (QOL) as affected by atopic dermatitis. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Time Frame: Baseline (Day 1) , Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Score on a Scale | -6.77 (0.497) [lower limit 0.497] | -10.75 (0.476) [lower limit 0.476] | -10.89 (0.469) [lower limit 0.469]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -4.11, 95% CI 2-sided [-5.434 to -2.796]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -3.98, 95% CI 2-sided [-5.298 to -2.657]

17. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurements Information Systems (PROMIS) Pediatric Anxiety Short Form Scale Total Score at Week 16
Description: PROMIS Anxiety instrument measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), & somatic symptoms related to arousal (racing heart, dizziness). Each question has 5 response options ranging in value from 1-5 (1=Never, 2=Almost never, 3=Sometimes, 4=Often, 5=Almost Always). Total raw score calculated using sum of response values: for 8-item form, lowest possible is 8 & highest possible is 40; For 6-item form: lowest possible is 6; highest possible is 30. Higher score indicates greater severity of symptoms.
Time Frame: Baseline (Day 1), Week 16
Population: The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Score on a Scale | -10.17 (0.912) [lower limit 0.912] | -13.19 (0.861) [lower limit 0.861] | -13.54 (0.860) [lower limit 0.860]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0061, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -3.37, 95% CI 2-sided [-5.779 to -0.962]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0133, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -3.02, 95% CI 2-sided [-5.414 to -0.629]

18. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurements Information Systems (PROMIS) Pediatric Depressive Symptoms Short Form Scale Score at Week 16
Description: PROMIS Depression instrument assesses self-reported negative mood (sadness/guilt), views of self (self-criticism/worthlessness) & social cognition (loneliness/interpersonal alienation), & decreased positive affect & engagement (loss of interest/meaning/purpose). Each question has 5 response options with values from 1-5 (1=Never, 2=Almost never, 3=Sometimes, 4=Often, 5=Almost Always). Total raw score is the sum of response values. For 8-item form, lowest possible is 8, highest is 40; for 6-item form, lowest possible is 6, highest is 30. Higher score indicates greater severity of symptoms.
Time Frame: Baseline (Day 1), Week 16
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Score on a Scale | -7.42 (0.848) [lower limit 0.848] | -12.84 (0.793) [lower limit 0.793] | -11.92 (0.790) [lower limit 0.790]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -4.5, 95% CI 2-sided [-6.734 to -2.272]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Square Mean Difference = -5.42, 95% CI 2-sided [-7.641 to -3.207]

19. Secondary Outcome: Percentage of Participants Having at Least One Skin Infection Treatment Emergent Adverse Event (TEAE) (Excluding Herpetic Infections) Through Week 16
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-subjects hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs. Percentage of participants having at least one skin infection TEAE (Excluding Herpetic Infections) through Week 16 were reported. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Time Frame: Baseline through Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percentage of Participants | 13.0 | 5.7 | 8.2
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.222, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage Differenece = -4.8, 95% CI 2-sided [-12.49 to 2.87]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0508, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Percentage Differenece = -7.3, 95% CI 2-sided [-14.51 to -0.03]

20. Secondary Outcome: Percentage of Participants Having at Least One Serious Treatment Emergent Adverse Event (TEAE) Through Week 16
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-participants hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Time Frame: Baseline (Day 1) through Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 122
Percentage of Participants | 1.6 | 1.6 | 0

21. Secondary Outcome: Proportion of Topical Corticosteroid (TCS) Medication-free Days From Baseline to Week 16
Description: Proportion of TCS medication-free days is calculated as the number of days that a participant used neither TCS/TCI nor system rescue therapy divided by the study days of each period. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Here "Number of participants analyzed" = number of participants who were evaluated for this specific endpoint.
Time Frame: Baseline (Day 1), Week 16
Measure: Mean (Standard Deviation); unit: Proportion of Days
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 123 | 122 | 121
Proportion of Days | 0.11 (0.185) [lower limit 0.185] | 0.20 (0.230) [lower limit 0.230] | 0.19 (0.207) [lower limit 0.207]

22. Secondary Outcome: Mean Weekly Dose of Topical Corticosteroid (TCS) in Grams for Low or Medium Potency TCS From Baseline to Week 16
Description: Mean weekly dose of TCS in grams for low or medium potency TCS from baseline to Week 16 were reported. The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Here "Number of participants analyzed" = number of participants who were evaluated for this specific endpoint.
Time Frame: Baseline (Day 1), Week 16
Measure: Least Squares Mean (Standard Error); unit: Grams
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
Number analyzed (Participants) | 120 | 120 | 120
Grams | 20.1 (1.37) [lower limit 1.37] | 15.0 (1.36) [lower limit 1.36] | 14.4 (1.38) [lower limit 1.38]
Statistical Analysis 1: Comparison: Placebo + TCS vs Dupilumab 100 mg or 200 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, ANOVA — The confidence interval (CI) with p-value was based on treatment difference (Dupilumab group vs placebo) of the LS mean percent change using ANOVA model with the treatment, randomization strata as fixed factors; Least Square Mean Difference = -5.7, 95% CI 2-sided [-9.49 to -1.96]
Statistical Analysis 2: Comparison: Placebo + TCS vs Dupilumab 300 mg Q4W + TCS; Test type: Superiority — A 2-sided hierarchical testing procedure was used for the primary and secondary endpoints in a pre-specified order. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level; p = 0.0082, ANOVA — [p-value comment as in outcome 22, analysis 1]; Least Square Mean Difference = -5.1, 95% CI 2-sided [-8.8 to -1.31]

ADVERSE EVENTS:
Time Frame: Reported AEs are treatment-emergent adverse events which were collected for both the 16-week treatment period and the follow-up period for as long as 12 weeks.
Description: The safety analysis set (SAF) includes all randomized subjects who received at least one injection of study drug and were analyzed as treated. Treatment compliance/administration and all clinical safety variables were summarized based on the SAF.
Arm/Group | Placebo + TCS | Dupilumab 300 mg Q4W + TCS | Dupilumab 100 mg or 200 mg Q2W + TCS
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120 | 0/122
Serious Adverse Events (participants affected / at risk) | 2/120 | 3/120 | 0/122
Other Adverse Events (participants affected / at risk) | 57/120 | 47/120 | 50/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + TCS (N=120) | Dupilumab 300 mg Q4W + TCS (N=120) | Dupilumab 100 mg or 200 mg Q2W + TCS (N=122)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + TCS (N=120) | Dupilumab 300 mg Q4W + TCS (N=120) | Dupilumab 100 mg or 200 mg Q2W + TCS (N=122)
Vomiting (Gastrointestinal disorders) | 8 (9) | 6 (7) | 6 (8)
Injection site erythema (General disorders) | 2 (3) | 5 (5) | 7 (9)
Conjunctivitis (Infections and infestations) | 3 (3) | 5 (5) | 7 (8)
Nasopharyngitis (Infections and infestations) | 8 (11) | 15 (16) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 14 (19) | 12 (16)
Viral upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 10 (11) | 6 (7) | 7 (10)
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 3 (3) | 5 (5)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 17 (25) | 8 (12) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT03345914/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03345914/SAP_001.pdf